CLINICAL TRIAL: NCT05216172
Title: AZD1656 in Transplantation With Diabetes tO PromoTe Immune TOleraNce
Acronym: ADOPTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 252155
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Type 2 Diabetes; Diabetes Mellitus, Type 2; Renal Transplant; Kidney Transplant; Complications; End Stage Renal Disease
Keywords: Type 2 Diabetes Mellitus; Diabetes Mellitus; Renal transplantation; Regulatory T cells; AZD1656
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Kidney Failure, Chronic; Diabetes Mellitus | interventions — AZD1656

STUDY DESIGN:
Intervention Model Description: Single site, placebo controlled, double blind randomised clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double blind placebo study: both the patient and the study team will be blinded to the treatment intervention.
  Pharmacy staff who dispense the study medication will not be blinded, nor will Sponsor Office staff responsible for reporting unblinded SUSAR reports to the MHRA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD1656 (Experimental): AZD1656 100mg BD for 3 months
  Interventions: Drug: AZD1656
- placebo (Placebo Comparator): placebo 100mg BD for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1656 — active drug
  Arms: AZD1656
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
AZD1656 in Transplantation with Diabetes tO PromoTe Immune TOleraNce: a single site, placebo-controlled, double-blind randomised clinical trial of AZD1656 in renal transplant patients with Type 2 diabetes

DETAILED DESCRIPTION:
Transplant recipients with pre-existing Type 2 diabetes frequently experience a deterioration in glycaemic control in the early post-transplant period, largely due to the significant immunosuppression burden at this stage. Elevated glucose profiles have been associated with poorer graft outcomes. The glucokinase activator AZD1656 has been shown to be a potent anti diabetic medication and safe in patients with T2DM, including those with chronic kidney disease. Recent data has shown that glucokinase activation increases regulatory T cell (Treg) migration and trafficking. The investigators propose to study the safety and efficacy of AZD1656 in optimising the glycaemic control and in stimulating Treg migration to the transplant kidney in a population of renal transplant patients with pre-existing T2DM.

ADOPTION is a single site, placebo-controlled, double-blind randomised clinical trial of AZD1656 in patients with Type 2 diabetes who have received a new renal transplant. Eligible, consented patients are randomised to a 3 month course of either active drug or placebo within 24 hours of transplantation. Clinical and laboratory data will be collected and assessed at baseline and throughout their participation in the study. The study plans to enrol 50 patients. There are no interim analyses planned. The primary endpoint will be the mean change in peripheral Tregs between baseline and 3 months as analysed by flow cytometry.

Ethical approval was obtained from the East of England - Cambridge East Ethics Committee (REC 19/EE/0209) prior to commencing the study. All study-related data will be used by the Sponsor in accordance with local data protection law. Results of the trial will be submitted for publication in a peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

1. Females or males aged 18 years and above
2. Having undergone renal transplantation at the Royal London Hospital within the previous 24 hours
3. A pre-transplant diagnosis of Type 2 diabetes
4. Provision of written, informed consent prior to any study specific procedures
5. In women of childbearing potential* documentation of a negative pregnancy test during admission for renal transplant.

   * Women of childbearing potential are defined as women following menarche until becoming post-menopausal, unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A post-menopausal state is defined as the absence of menses for 12 months without an alternative medical cause.

Exclusion Criteria:

1. Unable to consent
2. Known allergy/intolerance to AZD1656
3. Pregnant or breastfeeding women
4. Planning on becoming pregnant/unwilling to use highly effective contraception* during the 3 month treatment period and for 2 weeks afterwards (i) In the case of men with sexual partners who are women of childbearing potential: refusal to wear a condom and female partner planning on becoming pregnant/unwilling to use highly effective contraception* during the 3 month treatment period and for 2 weeks afterwards
5. Clinically significant history of abnormal physical and/or mental health as judged by the investigator other than conditions related to chronic kidney disease
6. Current or planned use of strong inhibitors of CYP2C8
7. Participation in an investigational drug trial in the 3 months prior to administration of the initial dose of study drug

   * Highly effective contraception methods are defined as those that can achieve a failure rate of <1% per year when used correctly and consistently. These include:

     * Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation - either oral, transvaginal or transdermal
     * Progestogen-only hormonal contraception associated with inhibition of ovulation - either oral, injectable or implantable
     * Intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
     * Bilateral tubal occlusion
     * Vasectomised partner - provided that the partner is the sole sexual partner of the participant and that the vasectomised partner has received medical assessment of surgical success

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2022-09-11 (Actual); Study Completion 2022-09-11 (Actual)

PRIMARY OUTCOMES:
peripheral regulatory T cells | 14 weeks
  Change in mean peripheral Treg cell number between baseline and 3 months measured using flow cytometry analysis (FACS) in AZD1656 and placebo arms

SECONDARY OUTCOMES:
regulatory T cells in renal transplant | 3 months
  Histological staining for Treg cells in renal biopsy tissue between baseline and 3 month protocol biopsy
delayed graft function | 1 week
  Incidence of delayed graft function, defined as the need for dialysis within 1 week post-transplant
glycemic control: HbA1c | 3 months
  Diabetic control between baseline and month 3 using change in HbA1c measurement
number of participants with increase or decrease in concurrent anti-diabetic medication | 3 months
  Dose of other anti-diabetic medication between baseline and month 3 (descriptive)
incidence of treatment emergent adverse events | 3 months
  safety endpoints including hypoglycaemic episodes
change in HOMA-IR measurement between baseline and month 3 | 3 months
  Insulin resistance: HOMA IR measurement at month 3
kidney transplant function | 3 months
  Graft function: (eGFR) at month 3
kidney transplant rejection | 3 months
  Episodes of acute rejection (defined as biopsy proven acute rejection)
incidence of treatment emergent adverse events (with particular reference to episodes of infection) | 3 months
  Episodes of opportunistic infections: bacterial and viral (descriptive)

OTHER OUTCOMES:
Comparison of patient and placebo group at 1 year post transplant: number of participants experiencing episodes of infection, rejection; comparison of renal function and diabetic control | 1 year
  12-month graft function (eGFR) and diabetic control (HbA1c; medication review) to assess legacy effect
T cell profile | 3 months
  Differences in other peripheral T cell populations, measured by FACS analysis
regulatory T cells in renal transplant: biopsy for cause | 3 months
  Histological staining for Treg cells in any renal biopsy taken for clinical indications between baseline and month 3 protocol biopsy
regulatory T cells: functional assay | 3 months
  Differences in the functional phenotype of the Treg cells

CONTACTS AND LOCATIONS:
Overall Officials: Kieran McCafferty, M.B., B.Chir, Principal Investigator — Barts Health NHS Trust; Queen Mary University London
Locations (1):
- Royal London Hospital Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in any published article, after de-identification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
  The data may be used for individual participant data meta-analysis.
  Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at [email corresponding author??]

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT05216172/Prot_SAP_000.pdf